CLINICAL TRIAL: NCT00443209
Title: A Multicenter, Double-Blind, Active-Controlled, Parallel Group Study to Examine the Safety, Tolerability and Efficacy of Oral MK-0974 for the Long Term Treatment of Acute Migraine With or Without Aura
Brief Title: Telcagepant (MK-0974) Long-Term Safety Study in Adult Participants With Acute Migraine (MK-0974-012)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0974-012; MK-0974-012 (Other: Merck Protocol Number); 2006_524 (Other: Telerx Study Number)
Record Dates: First submitted 2007-02-28; First posted 2007-03-05 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — telcagepant; rizatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telcagepant 280 mg/300 mg (Experimental): Participants receive telcagepant 300 mg soft gel capsules or telcagepant 280 mg tablets, administered orally as a single dose at onset of migraine. If still experiencing a migraine 2 hours after the first dose of telcagepant, participants may take an optional second dose of study drug or non-study rescue medication. Participants may take up to 16 doses (for treatment of up to 8 migraines) of telcagepant per month for up to 18 months.
  Interventions: Drug: Telcagepant 300 mg soft gel capsules; Drug: Telcagepant 280 mg tablets; Drug: Placebo to rizatriptan tablets
- Rizatriptan 10 mg (Active Comparator): Participants receive rizatriptan tablets, administered orally as a single dose at onset of migraine. If still experiencing a migraine 2 hours after the first dose of rizatriptan, participants may take an optional second dose of study drug or non-study rescue medication. Participants may take up to 16 doses (for treatment of up to 8 migraines) of rizatriptan per month for up to 18 months.
  Interventions: Drug: Rizatriptan 10 mg tablets; Drug: Placebo to telcagepant capsules; Drug: Placebo to telcagepant tablets

INTERVENTIONS:
Drug: Telcagepant 300 mg soft gel capsules — One capsule taken orally at onset of migraine
  Arms: Telcagepant 280 mg/300 mg
Drug: Telcagepant 280 mg tablets — One tablet taken orally at onset of migraine
  Arms: Telcagepant 280 mg/300 mg
Drug: Rizatriptan 10 mg tablets — One tablet taken orally at onset of migraine
  Arms: Rizatriptan 10 mg
Drug: Placebo to telcagepant capsules — One capsule taken orally at onset of migraine
  Arms: Rizatriptan 10 mg
Drug: Placebo to telcagepant tablets — One tablet taken orally at onset of migraine
  Arms: Rizatriptan 10 mg
Drug: Placebo to rizatriptan tablets — One tablet taken orally at onset of migraine
  Arms: Telcagepant 280 mg/300 mg

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of telcagepant (MK-0974) in the long-term treatment of acute migraine in adult participants. The primary hypothesis of this study is that telcagepant is well tolerated in the long-term treatment of acute migraine in adult participants.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 year history of migraine (with or without aura)
* Females of child bearing potential must use acceptable contraception throughout trial
* In general good health based on screening assessment

Exclusion Criteria:

* Pregnant/breast-feeding (or is a female expecting to conceive during study period)
* History or evidence of stroke/transient ischemic attacks, heart disease, coronary artery vasospasm, other significant underlying cardiovascular diseases, uncontrolled hypertension (high blood pressure), uncontrolled diabetes, or human immunodeficiency virus (HIV) disease
* Major depression, other pain syndromes that might interfere with study assessments, psychiatric conditions, dementia, or significant neurological disorders (other than migraine)
* History of gastric, or small intestinal surgery, or has a disease that causes malabsorption
* History of cancer within the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1068 (Actual)
Dates: Start 2007-02-21 (Actual); Primary Completion 2009-01-22 (Actual); Study Completion 2009-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Connor KM, Aurora SK, Loeys T, Ashina M, Jones C, Giezek H, Massaad R, Williams-Diaz A, Lines C, Ho TW. Long-term tolerability of telcagepant for acute treatment of migraine in a randomized trial. Headache. 2011 Jan;51(1):73-84. doi: 10.1111/j.1526-4610.2010.01799.x. Epub 2010 Nov 10. PMID 21070230
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0974-012&kw=0974-012&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The trial was considered to have achieved completion as defined by the treatment of 100 participants for 12 months.
Period: Months 1 to 12 Treatment Period
Arm/Group | Telcagepant 280 mg/300 mg | Rizatriptan 10 mg
Started | 712 | 356
Treated | 641 | 313
Completed | 367 (Trial terminated used for participants not completing 12 months of treatment due to trial completion) | 202 (Trial terminated used for participants not completing 12 months of treatment due to trial completion)
Not Completed | 345 | 154
Not completed — Adverse Event | 22 | 11
Not completed — Protocol Violation | 14 | 7
Not completed — Lack of Efficacy | 50 | 11
Not completed — Lack of Qualifying Event | 1 | 1
Not completed — Lost to Follow-up | 36 | 15
Not completed — Physician Decision | 8 | 4
Not completed — Pregnancy | 3 | 4
Not completed — Trial Terminated | 43 | 23
Not completed — Withdrawal by Subject | 95 | 34
Not completed — Missing | 2 | 1
Not completed — Not Treated | 71 | 43
Period: Months 13 to 18 Treatment Period
Arm/Group | Telcagepant 280 mg/300 mg | Rizatriptan 10 mg
Started | 186 (The Months 13 to 18 Treatment Period.was optional. 181 participants chose not to continue.) | 86 (The Months 13 to 18 Treatment Period was optional. 116 participants chose not to continue.)
Completed | 87 (Trial terminated used for participants not completing 18 months of treatment due to trial completion) | 39 (Trial terminated used for participants not completing 18 months of treatment due to trial completion)
Not Completed | 99 | 47
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Trial Terminated | 87 | 43
Not completed — Withdrawal by Subject | 7 | 2

BASELINE CHARACTERISTICS:
Population: Baseline Analyis Population consisted of All Treated Participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Telcagepant 280 mg/300 mg | Rizatriptan 10 mg | Total
Number analyzed (Participants) | 641 | 313 | 954
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.5 (10.9) | 41.9 (11.1) | 42.3 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 502 | 237 | 739
  Male | 139 | 76 | 215

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With At Least One Triptan-Related Adverse Experience (AE)
Description: Triptan-related AEs are defined as: chest pain, chest tightness, asthenia, paraesthesia, dysaesthesia or hyperaesthesia. Participants were monitored for triptan-related AEs for 14 days after any dose of study drug.
Time Frame: Within 14 days of any dose of study drug (Up to 18.5 months)
Population: The All-Patients-As-Treated (APAT) population consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Telcagepant 280 mg/300 mg | Rizatriptan 10 mg
Number analyzed (Participants) | 641 | 313
Percentage of Participants | 5.0 | 11.2
Statistical Analysis 1: Comparison: Telcagepant 280 mg/300 mg vs Rizatriptan 10 mg; Test type: Superiority or Other; p < 0.001, Miettenen and Nurminen method; Treatment Difference = -6.2, 95% CI 2-sided [-10.4 to -2.6] — Treatment Difference was compared using the Miettinen and Nurminen (MN) method

2. Primary Outcome: Percentage of Participants With At Least One Clinical AE
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the study product, is also an AE. A clinical AE was an AE reported as a result of a clinical examination. Participants were monitored for clinical AEs for 14 days after any dose of study drug.
Time Frame: Within 14 days of any dose of study drug (Up to 18.5 months)
Population: The APAT population consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Telcagepant 280 mg/300 mg | Rizatriptan 10 mg
Number analyzed (Participants) | 641 | 313
Percentage of Participants | 58.7 | 63.9
Statistical Analysis 1: Comparison: Telcagepant 280 mg/300 mg vs Rizatriptan 10 mg; Test type: Superiority or Other; Treatment Difference = -5.2, 95% CI 2-sided [-11.7 to 1.4] — Treatment Difference was compared using the MN method

3. Primary Outcome: Percentage of Participants With At Least One Laboratory AE
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the study product, is also an AE. A laboratory AE was an AE reported as a result of a laboratory assessment or test. Participants were monitored for laboratory AEs for 14 days after any dose of study drug.
Time Frame: Within 14 days of any dose of study drug (Up to 18.5 months)
Population: The APAT population consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Telcagepant 280 mg/300 mg | Rizatriptan 10 mg
Number analyzed (Participants) | 641 | 313
Percentage of Participants | 1.9 | 1.6
Statistical Analysis 1: Comparison: Telcagepant 280 mg/300 mg vs Rizatriptan 10 mg; Test type: Superiority or Other; Treatment Difference = 0.3, 95% CI 2-sided [-2.0 to 2.0] — Treatment Difference was compared using the MN method

4. Primary Outcome: Percentage of Participants With At Least One Vital Sign Measurement Outside Predefined Limits of Change
Description: Predefined limits of change were established for vital sign measurements: Systolic Blood Pressure (>=180 mm Hg and 20 mm Hg increase OR <=90 mm Hg and 20 mm Hg decrease), Diastolic Blood Pressure (>=105 mm Hg and 15 mm Hg increase OR <=50 mm Hg and 15 mm Hg decrease), Pulse (>=120 beats per minute [bpm] and 15 bpm increase OR <=50 bpm and 15 bpm decrease), Body Temperature (>38º C [oral equivalent]) and Respiratory Rate (>25 or increase of 10 OR <5 or decrease of 10 [per minute]). Participants were monitored for vital sign measurements outside predefined limits of change for 14 days after any dose of study drug.
Time Frame: Within 14 days of any dose of study drug (Up to 18.5 months)
Population: The APAT population consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Telcagepant 280 mg/300 mg | Rizatriptan 10 mg
Number analyzed (Participants) | 641 | 313
Percentage of Participants
  Systolic Blood Pressure Increase | 0.2 | 0.3
  Systolic Blood Pressure Decrease | 1.4 | 1.3
  Diastolic Blood Pressure Increase | 0.3 | 0.6
  Diastolic Blood Pressure Decrease | 1.1 | 1.0
  Pulse Increase | 0.0 | 0.0
  Pulse Decrease | 0.6 | 1.6
  Body Temperature Increase | 0.3 | 0.3
  Respiratory Rate Increase or Decrease | 0.8 | 0.6

5. Secondary Outcome: Percentage of Participant Migraine Attacks With Pain Freedom (PF) at 2 Hours Post-Dose
Description: Participants were asked to rate their migraine headache severity with ratings of 0=No pain, 1=Mild pain, 2=Moderate pain, and 3=Severe pain. PF at 2 hours post-dose is defined as a decrease from mild, moderate or severe migraine headache (Grade 1, 2, or 3) at baseline to no pain (Grade 0) 2 hours post-dose.
Time Frame: 2 hours post-dose (Up to 18 months)
Population: The Full Analysis Set (FAS) population consisted of all participants who were randomized and reported at least one treated migraine attack with at least one post-treatment efficacy evaluation.
Measure: Mean (Standard Deviation); unit: Percentage of Migraine Attacks
Arm/Group | Telcagepant 280 mg/300 mg | Rizatriptan 10 mg
Number analyzed (Participants) | 592 | 294
Percentage of Migraine Attacks | 38.9 (29.5) | 47.5 (29.7)
Statistical Analysis 1: Comparison: Telcagepant 280 mg/300 mg vs Rizatriptan 10 mg; Test type: Superiority or Other; Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.45 to 0.75] — Based on mixed logistic regression model with a fixed effect term for treatment, baseline pain severity and a random effect term for participant, with the random effect following a normal distribution. An odds ratio >1 is in favor of telcagepant

ADVERSE EVENTS:
Time Frame: Up to 14 days after any dose of study drug (Up to 18.5 months)
Description: The population consisted of all participants who received at least one dose of study drug.
Arm/Group | Telcagepant 280 mg/300 mg | Rizatriptan 10 mg
Serious Adverse Events (participants affected / at risk) | 12/641 | 6/313
Other Adverse Events (participants affected / at risk) | 187/641 | 127/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telcagepant 280 mg/300 mg (N=641) | Rizatriptan 10 mg (N=313)
Vertigo (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1 | 0
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sqamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telcagepant 280 mg/300 mg (N=641) | Rizatriptan 10 mg (N=313)
Dry mouth (Gastrointestinal disorders) | 62 | 43
Nausea (Gastrointestinal disorders) | 58 | 20
Asthenia (General disorders) | 14 | 16
Fatigue (General disorders) | 31 | 32
Upper respiratory tract infection (Infections and infestations) | 17 | 16
Dizziness (Nervous system disorders) | 57 | 32
Somnolence (Nervous system disorders) | 59 | 52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.